CLINICAL TRIAL: NCT02811861
Title: A Multicenter, Open-label, Randomized, Phase 3 Trial to Compare the Efficacy and Safety of Lenvatinib in Combination With Everolimus or Pembrolizumab Versus Sunitinib Alone in First-Line Treatment of Subjects With Advanced Renal Cell Carcinoma (CLEAR)
Brief Title: Lenvatinib/Everolimus or Lenvatinib/Pembrolizumab Versus Sunitinib Alone as Treatment of Advanced Renal Cell Carcinoma
Acronym: CLEAR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7080-G000-307; KEYNOTE-581 (Other: Merck); 2016-000916-14 (EudraCT Number)
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Results first posted 2021-09-24 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma (RCC); Lenvatinib; First-line RCC; Treatment-naive RCC; Everolimus; Pembrolizumab; Sunitinib; Phase 3 RCC; Phase 3 first-line RCC; Phase 3 treatment-naive RCC
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — lenvatinib; Everolimus; pembrolizumab; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lenvatinib 18 mg plus Everolimus 5 mg (Experimental): Lenvatinib 18 milligrams (mg) administered orally, once daily, plus everolimus 5 mg administered orally, once daily in each 21-day cycle.
  Interventions: Drug: Lenvatinib; Drug: Everolimus
- Lenvatinib 20 mg plus Pembrolizumab 200 mg (Experimental): Lenvatinib 20 mg administered orally, once daily, in each 21-day cycle plus pembrolizumab 200 mg administered intravenously (IV), every 3 weeks on Day 1 of each 21-day cycle.
  Interventions: Drug: Lenvatinib; Drug: Pembrolizumab
- Sunitinib 50 mg (Active Comparator): Sunitinib 50 mg administered orally, once daily, on a schedule of 4 weeks on treatment followed by 2 weeks off treatment in each 21-day cycle.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Lenvatinib
  Arms: Lenvatinib 18 mg plus Everolimus 5 mg; Lenvatinib 20 mg plus Pembrolizumab 200 mg
Drug: Everolimus
  Arms: Lenvatinib 18 mg plus Everolimus 5 mg
Drug: Pembrolizumab
  Arms: Lenvatinib 20 mg plus Pembrolizumab 200 mg
Drug: Sunitinib
  Arms: Sunitinib 50 mg

SUMMARY:
The primary purpose of the study is to demonstrate that lenvatinib in combination with everolimus (Arm A) or pembrolizumab (Arm B) is superior compared to sunitinib alone (Arm C) in improving progression-free survival (PFS) (by independent imaging review [IIR] using Response Evaluation Criteria in Solid Tumors [RECIST 1.1]) as first-line treatment in participants with advanced renal cell carcinoma (RCC).

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological confirmation of RCC with a clear-cell component (original tissue diagnosis of RCC is acceptable).
2. Documented evidence of advanced RCC.
3. At least 1 measurable target lesion according to RECIST 1.1 meeting the following criteria:

   * Lymph node (LN) lesion that measures at least 1 dimension as greater than or equal to (>=) 1.5 cm in the short axis
   * Lymph node (LN) lesion that measures at least 1 dimension as greater than or equal to (>=) 1.5 centimeter (cm) in the short axis
   * Non-nodal lesion that measures greater than or equal to (>=) 1.0 cm in the longest diameter
   * The lesion is suitable for repeat measurement using computerized tomography/magnetic resonance imaging (CT/MRI). Lesions that have had external beam radiotherapy (EBRT) or locoregional therapy must show radiographic evidence of disease progression based on RECIST 1.1 to be deemed a target lesion.

3.Karnofsky Performance Status (KPS) of >=70 4.Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP less than or equal (<=) 150/90 millimeter of mercury (mmHg) at Screening and no change in antihypertensive medications within 1 week prior to Cycle 1/Day 1 (C1/D1) 5.Adequate renal function defined as creatinine <=1.5*upper limit of normal (ULN); or for participants with creatinine greater than (>) 1.5*ULN, the calculated creatinine clearance >=30 milliliters per minute (mL/min) (per the Cockcroft-Gault formula) is acceptable.

6.Adequate bone marrow function defined by:

* Absolute neutrophil count (ANC) >=1500/cubic millimeter (mm^3)
* Platelets >=100,000/mm^3
* Hemoglobin >=9 grams per deciliter (g/dL) NOTE: Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within the previous 2 weeks.

  7.Adequate blood coagulation function defined by International Normalized ratio (INR) <=1.5 unless participant is receiving anticoagulant therapy, as long as INR is within therapeutic range of intended use of anticoagulants.

  8.Adequate liver function defined by:
* Total bilirubin <=1.5*ULN except for unconjugated hyperbilirubinemia of Gilbert's syndrome.
* Alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) <=3*ULN (in the case of liver metastases <=5*ULN), unless there are bone metastases. Participants with ALP values >3*ULN and known to have bone metastases can be included.

  9.Provide written informed consent. 10.Willing and able to comply with all aspects of the protocol.

Exclusion Criteria:

1. Participants who have received any systemic anticancer therapy for RCC, including anti-vascular endothelial growth factor (VEGF) therapy, or any systemic investigational anticancer agent. Prior adjuvant treatment with an investigational anticancer agent is not allowed unless the investigator can provide evidence of participant's randomization to placebo arm.
2. Participants with central nervous system (CNS) metastases are not eligible, unless they have completed local therapy (example, whole brain radiation therapy (WBRT), surgery or radiosurgery) and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment in this study. Any signs (example, radiologic) or symptoms of CNS metastases must be stable for at least 4 weeks before starting study treatment
3. Active malignancy (except for RCC, definitively treated basal or squamous cell carcinoma of the skin, and carcinoma in-situ of the cervix or bladder) within the past 24 months. Participants with history of localized & low risk prostate cancer are allowed in the study if they were treated with curative intent and there is no prostate specific antigen (PSA) recurrence within the past 5 years
4. Prior radiation therapy within 21 days prior to start of study treatment with the exception of palliative radiotherapy to bone lesions, which is allowed if completed 2 weeks prior to study treatment start
5. Participants who are using other investigational agents or who had received investigational drugs <=4 weeks prior to study treatment start.
6. Received a live vaccine within 30 days of planned start of study treatment (Cycle 1/Day 1). Examples of live vaccines include, but are not limited to, measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (example, FluMist®) are live attenuated vaccines and are not allowed.
7. Participants with proteinuria >1+ on urine dipstick testing will undergo 24-h urine collection for quantitative assessment of proteinuria. Participants with urine protein >=1 g/24 h will be ineligible
8. Fasting total cholesterol >300 milligram per deciliter (mg/dL) (or ˃7.75 millimole per liter (mmol/L)) and/or fasting triglycerides level ˃2.5 x upper limit of normal (ULN). Note: these participants can be included after initiation or adjustment of lipid-lowering medication
9. Uncontrolled diabetes as defined by fasting glucose >1.5 times the ULN. Note: these participants can be included after initiation or adjustment of glucose-lowering medication
10. Prolongation of corrected QT (QTc) interval to >480 milliseconds (ms)
11. Participants who have not recovered adequately from any toxicity and/or complications from major surgery prior to starting therapy.
12. Gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib, everolimus, and/or sunitinib.
13. Bleeding or thrombotic disorders or participants at risk for severe hemorrhage. The degree of tumor invasion/infiltration of major blood vessels should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy
14. Clinically significant hemoptysis or tumor bleeding within 2 weeks prior to the first dose of study drug
15. Significant cardiovascular impairment within 12 months of the first dose of study drug: history of congestive heart failure greater than New York Heart Association Class II, unstable angina, myocardial infarction, cerebrovascular accident, or cardiac arrhythmia associated with hemodynamic instability. The following is also excluded: left ventricular ejection fraction (LVEF) below the institutional normal range as determined by multiple-gated acquisition MUGA scan or echocardiogram
16. Active infection (any infection requiring systemic treatment)
17. Participants known to be positive for Human Immunodeficiency Virus (HIV).
18. Known active Hepatitis B (example, Hepatitis B surface antigen (HBsAg) reactive) or Hepatitis C (example, hepatitis C virus ribonucleic acid (HCV RNA) [qualitative] is detected)
19. Known history of, or any evidence of, interstitial lung disease
20. Has a history of (non-infectious) pneumonitis that required steroids, or current pneumonitis
21. Participants with a diagnosis of immunodeficiency or who are receiving chronic systemic steroid therapy (doses exceeding 10 mg/day of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment. Physiologic doses of corticosteroids (up to 10 mg/day of prednisone or equivalent) may be used during the study
22. Active autoimmune disease (with the exception of psoriasis) that has required systemic treatment in the past 2 years (that is, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (example, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
23. Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [ß-hCG] (or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 IU/L or equivalent units of ß-hCG [or hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
24. Females of childbearing potential who:

    * Do not agree to use a highly effective method of contraception for the entire study period and for 120 days after study discontinuation, that is:
    * total abstinence (if it is their preferred and usual lifestyle)
    * an intrauterine device (IUD) or hormone-releasing system (IUS)
    * a contraceptive implant
    * an oral contraceptive (with additional barrier method) OR
    * Do not have a vasectomized partner with confirmed azoospermia. For sites outside of the EU, it is permissible that if a highly effective method of contraception is not appropriate or acceptable to the participant, then the participant must agree to use a medically acceptable method of contraception, that is, double barrier methods of contraception such as condom plus diaphragm or cervical/vault cap with spermicide.
25. Males who have not had a successful vasectomy (confirmed azoospermia) and do not agree to use condom + spermicide OR have a female partner who does not meet the criteria above (that is, is of childbearing potential and not practicing highly effective contraception throughout the study period), starting with the first dose of study therapy through 120 days after the last dose of study therapy, unless sexually abstinent. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the participant.
26. Known intolerance to any of the study drugs (or any of the excipients)
27. Participant has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1069 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2026-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Locations (183):
- United States (35):
  - Stanford School of Medicine, Stanford, California
  - Boca Raton Community Hospital, Boca Raton, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - University of Miami, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Florida Cancer Specialists ( North Region), St. Petersburg, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Joliet Oncology - Hematology Associates, Joliet, Illinois
  - Healthcare Research Network III, LLC, Tinley Park, Illinois
  - Health Midwest Ventures Group, Inc d/b/a HCA MidAmerica Division, LLC, Overland Park, Kansas
  - Cotton-Oneil Clinical Research Center, Topeka, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Associates in Oncology & Hematology, PC, Bethesda, Maryland
  - Massachusetts General Hospital- MGH, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - GU Research Network, Omaha, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Hackensack Medical Center, Hackensack, New Jersey
  - Rosewell Park Cancer Institute, Buffalo, New York
  - Broome Oncology, Johnson City, New York
  - Weill Cornell Medical College New York Presbyterian Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Mission Hospital_ Cancer Care of Western North Carolina, Asheville, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - SCRI - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology, P.A., Dallas, Texas
  - Texas Oncology PA, Fort Worth, Texas
  - Texas Oncology PA - McAllen, McAllen, Texas
  - Texas Oncology PA - Paris, Paris, Texas
  - USOR Texas Oncology, The Woodlands, Texas
  - Texas Oncology PA - Tyler, Tyler, Texas
- Australia (6):
  - Box Hill Hospital, Box Hill, Victoria
  - Austin Health, Heidelberg, Victoria
  - Royal Hobart Hospital, Hobart
  - Macquarie University Hospital, Macquarie Park
  - ICON Cancer Foundation, South Brisbane
  - Sunshine Hospital, St Albans
- Austria (3):
  - Medizinische Universitat Innsbruck, Innsbruck
  - Krankenhaus der barmherzigen Schwestern Linz, Linz
  - AKH - Medizinische Universität Wien, Vienna
- Belgium (7):
  - O.L.V Ziekenhuis, Aalst
  - ZNA Middelheim, Antwerp
  - Imeldaziekenhuis, Bonheiden
  - Institut Jules Bordet, Brussels
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - Domaine Universitaire, Liège
  - GZA Ziekenhuizen - Campus Sint-Augustinus, Wilrijk
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency Vancouver Centre, Vancouver, British Columbia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - London Institute of Health Sciences, London, Ontario
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Research Institute - University of Toronto, Toronto, Ontario
  - Centre de santé et de services sociaux Champlain-Charles-Le Moyne, Greenfield Park, Quebec
- Czechia (6):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Olomouc, Neurologicka klinika, Olomouc
  - Fakultni nemocnice v Motole, Prague
  - Nemocnice Na Bulovce, Prague
  - Thomayerova nemocnice, Prague
- France (9):
  - ICO - Site Paul Papin, Angers, Maine Et Loire
  - Centre Georges François Leclerc, Dijon
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans
  - Centre Leon Berard - Centre regional de lutte contre le cancer Rhone-Alpes, Lyon
  - Institut Regional du Cancer de Montpellier, Montpellier
  - Hopital la Petie Salpetriere, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Boulevard du Professeur Jacques Monod, Saint-Herblain
  - CHU Strasbourg - Nouvel Hopital Civil, Strasbourg
- Germany (9):
  - EISAI Trial site 4, Stuttgart, Baden-Wurttemberg
  - EISAI Trial site 1, Tübingen, Baden-Wurttemberg
  - EISAI Trial site 7, München, Bavaria
  - EISAI Trial site 6, Frankfurt am Main, Hesse
  - EISAI Trial site 8, Hanover, Lower Saxony
  - EISAI Trial site 14, Greifswald, Mecklenburg-Vorpommern
  - EISAI Trial site 13, Münster, North Rhine-Westphalia
  - EISAI Trial site 2, Homburg/Saar, Saarland
  - EISAI Trial site 5, Berlin
- Greece (4):
  - General Hospital of Athens "Alexandra", Athens
  - University of Patras Medical School, Pátrai
  - General Hospital Papageorgiou, Thessaloniki
  - Interbalkan Hospital of Thessaloniki, Thessaloniki
- Ireland (4):
  - Cork University Hospital,Wilton, Cork
  - Adelaide and Meath Hospital Incorp The National Children's Hospital, Dublin
  - Beaumont Hospital, Dublin
  - University Hospital Galway, Galway
- Israel (6):
  - Assaf Harofeh Medical Center, Be’er Ya‘aqov
  - Rambam MC, Haifa
  - Sapir Medical Center, Meir Hospital, Kfar Saba
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (15):
  - Azienda Unità Sanitaria Locale- Ravenna, Faenza, Ravenna
  - Ospedale San Donato, Arezzo
  - Azienda Ospedaliera Universitaria Policlinico SantOrsola Malpighi, Bologna
  - Istituto Nazionale per la Ricerca sul Cancro di Genova, Genova
  - Presidio Ospedaliero Vito Fazzi, Lecce
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori - IRST, Meldola
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - A.O.U. Policlinico di Modena, Modena
  - Azienda Ospedaliera di Rilievo Nazionale A. Cardarelli, Napoli
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - I.R.C.S.S Fondazione Maugeri, Pavia
  - Azienda Ospedaliera Santa Maria Degli Angeli, Pordenone
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Universita Campus Bio-Medico di Roma, Rome
- Japan (26):
  - Facility #1, Aichi
  - Facility #1, Akita
  - Facility #1, Aomori
  - Facility #2, Chiba
  - Facility #1, Fukuoka
  - Facility #1, Hiroshima
  - Facility #1, Hokkaido
  - Facility #2, Hokkaido
  - Facility #1, Hyōgo
  - Facility #1, Kagawa
  - Facility #2, Kanagawa
  - Facility #3, Kanagawa
  - Facility #1, Nagasaki
  - Facility #1, Nara
  - Facility #1, Niigata
  - Facility #1, Okayama
  - Facility #1, Osaka
  - Facility #2, Osaka
  - Facility #1, Saitama
  - Facility #1, Tokushima
  - Facility #1, Tokyo
  - Facility #2, Tokyo
  - Facility #3, Tokyo
  - Facility #4, Tokyo
  - Facility #5, Tokyo
  - Facility #6, Tokyo
- Netherlands (3):
  - Antoni van Leeuwenhoek, Amsterdam
  - VU Medisch Centrum, Amsterdam
  - UMC Utrecht, Utrecht
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - SPWSZ w Szczecinie im. Marii Sklodowskiej-Curie, Szczecin
- Russia (7):
  - FSBSI Russian Oncological Scientific Center n.a. N.N. Blokhin - Department of Oncology, Moscow
  - FSBI "Moscow scientific research oncology institute n.a. P.A. Gertsen" of MoH of RF, Moscow
  - FSBSI Russian Oncological Scientific Center n.a. N.N. Blokhin - Department of Urology, Moscow
  - FBHI Privolzhskiy District Medical Centre FMBA of Russia, Nizhny Novgorod
  - SBHI of Novosibirsk region "Novosibirsk Regional Oncological Dispensary", Novosibirsk
  - FSBI "National Medical Research Radiological Center" of the MoH of the RF, Obninsk
  - BHI of Omsk region "Clinical Oncology Dispensary", Omsk
- South Korea (9):
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Asan Medical Center: Medical Oncology Department, Seoul
  - Asan Medical Center: Urology Department, Seoul
  - Department of Internal Medicine Division of Hematology/Oncology Cancer center 11F, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (15):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - ICO l'Hospitalet - Hospital Duran I Reynals, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario HM Madrid Sanchinarro, Madrid
  - MD Anderson Cancer Centre, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Virgen del Rocio, Seville
  - Oncologia, Valencia
- Inselspital - Universitaetsspital Bern, Bern, Switzerland
- United Kingdom (8):
  - Royal Bournemouth General Hospital, Bournemouth
  - Velindre Cancer Centre, Cardiff
  - Western General Hospital, Edinburgh
  - Beatson West Of Scotland Cancer Centre, Glasgow
  - St. James's University Hospital, Leeds
  - Guy's Hospital, London
  - Royal Free Hospital, London
  - Christie Hospital NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Fawsitt CG, Pan J, Orishaba P, Jackson CH, Thom H. Unanchored simulated treatment comparison on survival outcomes using parametric and Royston-Parmar models with application to lenvatinib plus pembrolizumab in renal cell carcinoma. BMC Med Res Methodol. 2025 Jan 30;25(1):26. doi: 10.1186/s12874-025-02480-x. PMID 39885377
- [Derived] Zheng H, Zhou J, Tong Y, Zhang J. Cost-Effectiveness Analysis of Lenvatinib plus Pembrolizumab or Everolimus as First-Line Treatment for Advanced Renal Cell Carcinoma. Clin Genitourin Cancer. 2025 Feb;23(1):102264. doi: 10.1016/j.clgc.2024.102264. Epub 2024 Nov 15. PMID 39642774
- [Derived] Motzer RJ, Choueiri TK, Hutson T, Young Rha S, Puente J, Lalani AA, Winquist E, Eto M, Basappa NS, Tannir NM, Vaishampayan U, Bjarnason GA, Oudard S, Grunwald V, Burgents J, Xie R, McKenzie J, Powles T. Characterization of Responses to Lenvatinib plus Pembrolizumab in Patients with Advanced Renal Cell Carcinoma at the Final Prespecified Survival Analysis of the Phase 3 CLEAR Study. Eur Urol. 2024 Jul;86(1):4-9. doi: 10.1016/j.eururo.2024.03.015. Epub 2024 Apr 6. PMID 38582713
- [Derived] Motzer RJ, Porta C, Eto M, Powles T, Grunwald V, Hutson TE, Alekseev B, Rha SY, Merchan J, Goh JC, Lalani AA, De Giorgi U, Melichar B, Hong SH, Gurney H, Mendez-Vidal MJ, Kopyltsov E, Tjulandin S, Gordoa TA, Kozlov V, Alyasova A, Winquist E, Maroto P, Kim M, Peer A, Procopio G, Takagi T, Wong S, Bedke J, Schmidinger M, Rodriguez-Lopez K, Burgents J, He C, Okpara CE, McKenzie J, Choueiri TK; CLEAR Trial Investigators. Lenvatinib Plus Pembrolizumab Versus Sunitinib in First-Line Treatment of Advanced Renal Cell Carcinoma: Final Prespecified Overall Survival Analysis of CLEAR, a Phase III Study. J Clin Oncol. 2024 Apr 10;42(11):1222-1228. doi: 10.1200/JCO.23.01569. Epub 2024 Jan 16. PMID 38227898
- [Derived] Grunwald V, Powles T, Eto M, Kopyltsov E, Rha SY, Porta C, Motzer R, Hutson TE, Mendez-Vidal MJ, Hong SH, Winquist E, Goh JC, Maroto P, Buchler T, Takagi T, Burgents JE, Perini R, He C, Okpara CE, McKenzie J, Choueiri TK. Phase 3 CLEAR study in patients with advanced renal cell carcinoma: outcomes in subgroups for the lenvatinib-plus-pembrolizumab and sunitinib arms. Front Oncol. 2023 Aug 16;13:1223282. doi: 10.3389/fonc.2023.1223282. eCollection 2023. PMID 37664025
- [Derived] Rha SY, Choueiri TK, Matveev VB, Alyasova A, Hong SH, Gordoa TA, Gurney H, Bjarnason GA, Buchler T, Pedrazzoli P, Takagi T, Park SH, Lee JL, Perini RF, He CS, McKenzie JA, Eto M. Efficacy and safety of lenvatinib plus pembrolizumab vs sunitinib in the East Asian subset of patients with advanced renal cell carcinoma from the CLEAR trial. Int J Cancer. 2023 Sep 15;153(6):1241-1250. doi: 10.1002/ijc.34608. Epub 2023 Jun 9. PMID 37294085
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Motzer R, George S, Merchan JR, Hutson TE, Song X, Perini RF, Xie R, Bapat U, Puente J. Characterization and Management of Adverse Reactions From the CLEAR Study in Advanced Renal Cell Carcinoma Treated With Lenvatinib Plus Pembrolizumab. Oncologist. 2023 Jun 2;28(6):501-509. doi: 10.1093/oncolo/oyac269. PMID 36866412
- [Derived] Choueiri TK, Eto M, Motzer R, De Giorgi U, Buchler T, Basappa NS, Mendez-Vidal MJ, Tjulandin S, Hoon Park S, Melichar B, Hutson T, Alemany C, McGregor B, Powles T, Grunwald V, Alekseev B, Rha SY, Kopyltsov E, Kapoor A, Alonso Gordoa T, Goh JC, Staehler M, Merchan JR, Xie R, Perini RF, Mody K, McKenzie J, Porta CG. Lenvatinib plus pembrolizumab versus sunitinib as first-line treatment of patients with advanced renal cell carcinoma (CLEAR): extended follow-up from the phase 3, randomised, open-label study. Lancet Oncol. 2023 Mar;24(3):228-238. doi: 10.1016/S1470-2045(23)00049-9. PMID 36858721
- [Derived] Motzer R, Porta C, Alekseev B, Rha SY, Choueiri TK, Mendez-Vidal MJ, Hong SH, Kapoor A, Goh JC, Eto M, Bennett L, Wang J, Pan JJ, Saretsky TL, Perini RF, He CS, Mody K, Cella D. Health-related quality-of-life outcomes in patients with advanced renal cell carcinoma treated with lenvatinib plus pembrolizumab or everolimus versus sunitinib (CLEAR): a randomised, phase 3 study. Lancet Oncol. 2022 Jun;23(6):768-780. doi: 10.1016/S1470-2045(22)00212-1. Epub 2022 Apr 27. PMID 35489363
- [Derived] Motzer R, Alekseev B, Rha SY, Porta C, Eto M, Powles T, Grunwald V, Hutson TE, Kopyltsov E, Mendez-Vidal MJ, Kozlov V, Alyasova A, Hong SH, Kapoor A, Alonso Gordoa T, Merchan JR, Winquist E, Maroto P, Goh JC, Kim M, Gurney H, Patel V, Peer A, Procopio G, Takagi T, Melichar B, Rolland F, De Giorgi U, Wong S, Bedke J, Schmidinger M, Dutcus CE, Smith AD, Dutta L, Mody K, Perini RF, Xing D, Choueiri TK; CLEAR Trial Investigators. Lenvatinib plus Pembrolizumab or Everolimus for Advanced Renal Cell Carcinoma. N Engl J Med. 2021 Apr 8;384(14):1289-1300. doi: 10.1056/NEJMoa2035716. Epub 2021 Feb 13. PMID 33616314
- [Derived] Hofmann F, Hwang EC, Lam TB, Bex A, Yuan Y, Marconi LS, Ljungberg B. Targeted therapy for metastatic renal cell carcinoma. Cochrane Database Syst Rev. 2020 Oct 14;10(10):CD012796. doi: 10.1002/14651858.CD012796.pub2. PMID 33058158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 181 investigative sites in Austria, Belgium, Canada, France, Germany, Greece, Ireland, Italy, Netherlands, Poland, Spain, Switzerland, United Kingdom of Great Britain and Northern Ireland, the United States of America, Australia, Czechia, Israel, Japan, Korea, Russian Federation, from 13 October 2016 to 28 August 2020 (date of data cutoff for the primary analysis of PFS and second interim analysis of Overall Survival).
Pre-assignment Details: A total of 1417 participants were screened, of which, 1069 were randomized. Of the 1069 randomized, 1047 participants were treated in the study.
Groups:
- Lenvatinib 18 mg Plus Everolimus 5 mg: Participants received lenvatinib 18 milligrams (mg) administered orally, once daily in each 21-day cycle, plus everolimus 5 mg administered orally, once daily in each 21-day cycle until participant had disease progression, development of unacceptable toxicity, participant request, withdrawal of consent.
- Lenvatinib 20 mg Plus Pembrolizumab 200 mg: Participants received lenvatinib 20 mg administered orally, once daily in each 21-day cycle, plus pembrolizumab 200 mg administered intravenously, every 3 weeks in each 21-day cycle until participant had disease progression, development of unacceptable toxicity, participant request, withdrawal of consent, completion of 35 treatments (approximately 2 years) with pembrolizumab, or sponsor termination of the study.
- Sunitinib 50 mg: Participants received sunitinib 50 mg administered orally, once daily, on a schedule of 4 weeks on treatment followed by 2 weeks off treatment until participant had disease progression, development of unacceptable toxicity, participant request, withdrawal of consent.
Period: Overall Study
Arm/Group | Lenvatinib 18 mg Plus Everolimus 5 mg | Lenvatinib 20 mg Plus Pembrolizumab 200 mg | Sunitinib 50 mg
Started | 357 | 355 | 357
Treated | 355 | 352 | 340
Completed | 0 | 0 | 0
Not Completed | 357 | 355 | 357
Not completed — Radiological Disease Progression | 123 | 97 | 174
Not completed — Clinical Disease Progression | 20 | 19 | 22
Not completed — Adverse Event | 63 | 60 | 41
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Subject Choice | 29 | 17 | 23
Not completed — Withdrawal by Subject | 4 | 4 | 9
Not completed — Other | 4 | 13 | 3
Not completed — Treatment Ongoing at Cutoff Date | 112 | 142 | 67
Not completed — Randomized but not treated | 2 | 3 | 17

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants regardless of the treatment actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenvatinib 18 mg Plus Everolimus 5 mg | Lenvatinib 20 mg Plus Pembrolizumab 200 mg | Sunitinib 50 mg | Total
Number analyzed (Participants) | 357 | 355 | 357 | 1069
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (10.86) | 62.3 (10.23) | 60.8 (9.96) | 61.7 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 100 | 82 | 273
  Male | 266 | 255 | 275 | 796
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 12 | 20 | 55
  Not Hispanic or Latino | 328 | 339 | 334 | 1001
  Unknown or Not Reported | 6 | 4 | 3 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 254 | 263 | 270 | 787
  Black or African American | 1 | 2 | 3 | 6
  Asian | 77 | 81 | 67 | 225
  American Indian or Alaskan Native | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Other | 7 | 4 | 7 | 18
  Missing | 16 | 5 | 10 | 31

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) by Independent Imaging Review (IIR)
Description: PFS assessed by IIR was defined as the time from the date of randomization to the date of the first documentation of progressive disease (PD) or death (whichever occurred first) using Response Evaluation Criteria in Solid Tumors (RECIST 1.1). PD was defined as at least a 20 percent (%) increase or 5 millimeter (mm) increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions. PFS was analyzed using Kaplan-Meier method.
Time Frame: From the date of randomization to the date of the first documentation of PD or date of death, whichever occurred first or up to data cutoff date 28 Aug 2020 (up to approximately 46 months)
Population: The FAS included all randomized participants regardless of the treatment actually received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib 18 mg Plus Everolimus 5 mg | Lenvatinib 20 mg Plus Pembrolizumab 200 mg | Sunitinib 50 mg
Number analyzed (Participants) | 357 | 355 | 357
months | 14.7 [11.1 to 16.7] | 23.9 [20.8 to 27.7] | 9.2 [6.0 to 11.0]
Statistical Analysis 1: Comparison: Lenvatinib 18 mg Plus Everolimus 5 mg vs Sunitinib 50 mg; Test type: Superiority; p < 0.0001, Stratified Log-rank Test; Hazard ratio is based on a Cox Proportional Hazards Model including treatment group as a factor; Stratified Hazard Ratio = 0.65, 95% CI 2-sided [0.53 to 0.80]
Statistical Analysis 2: Comparison: Lenvatinib 20 mg Plus Pembrolizumab 200 mg vs Sunitinib 50 mg; Test type: Superiority; p < 0.0001, Stratified Log-rank Test; Hazard ratio is based on a Cox Proportional Hazards Model including treatment group as a factor; Stratified Hazard Ratio = 0.39, 95% CI 2-sided [0.32 to 0.49]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the proportion of participants who had best overall response (BOR) of complete response (CR) or partial response (PR) as determined by IIR using RECIST 1.1. CR is defined as disappearance of all (targeted and non-target [NT]) lesions. All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to less than (<) 10mm. PR: defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. To be considered a BOR, all responses had to be confirmed no less than 4 weeks after the initial assessment of response. Data for this outcome measure will be reported after study completion (anticipated study completion date is March 2026).
Time Frame: Up to approximately 69 months
Reporting Status: Not Posted, anticipated posting 2027-03

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization to the date of death from any cause. Participants who were lost to follow-up and those who were alive at the data cutoff date were censored, either at the last date the participant was last known alive or at the data cutoff date, whichever occurred first. Data for this outcome measure will be reported after study completion (anticipated study completion date is March 2026).
Time Frame: Up to approximately 69 months
Reporting Status: Not Posted, anticipated posting 2027-03

4. Secondary Outcome: Number of Participants With At Least One Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAEs were defined as those adverse events (AEs) that occurred (or worsened, if present at Baseline) after the first dose of study drug through 30 days after the last dose of study drug.An AE was defined as any untoward medical occurrence in a participants or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. A SAE was defined as any AE if it resulted in death or life-threatening AE or required inpatient hospitalization or prolongation of existing hospitalization or resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions or was a congenital anomaly/birth defect. Data for this outcome measure will be reported after study completion (anticipated study completion date is March 2026).
Time Frame: Up to approximately 69 months
Reporting Status: Not Posted, anticipated posting 2027-03

5. Secondary Outcome: Number of Participants Who Discontinued Treatment Due to Toxicity
Description: Data for this outcome measure will be reported after study completion (anticipated study completion date is March 2026.
Time Frame: Up to approximately 69 months
Reporting Status: Not Posted, anticipated posting 2027-03

6. Secondary Outcome: Time to Treatment Failure Due to Toxicity
Description: Time to treatment failure due to toxicity is defined as time from the date of randomization to the date that a participant discontinued study treatment due to TEAEs. Data for this outcome measure will be reported after study completion (anticipated study completion date is March 2026).
Time Frame: Up to approximately 69 months
Reporting Status: Not Posted, anticipated posting 2027-03

7. Secondary Outcome: Health-Related Quality of Life (HRQoL) Assessed by Functional Assessment of Cancer Therapy Kidney Syndrome Index-Disease-Related Symptoms (FKSI-DRS) Scores
Description: The FKSI-DRS consisted of 9 items that experts and participants had indicated are important targets for the treatment of advanced kidney cancer, and that clinical experts had indicated are primarily disease-related, as opposed to treatment-related. Symptoms assessed on the FKSI-DRS included lack of energy, fatigue, weight loss, pain, bone pain, shortness of breath, cough, fever, or hematuria. Each item was scored on a 5-point Likert-type scale (0 = not at all; 4 = very much) where total score ranged from 0 (worst) to 36 (best), where higher scores correspond to better outcomes. Data for this outcome measure will be reported after study completion (anticipated study completion date is March 2026).
Time Frame: Up to approximately 69 months
Reporting Status: Not Posted, anticipated posting 2027-03

8. Secondary Outcome: HRQoL Assessed by European Organisation for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire C30 (QLQ-C30) Score
Description: EORTC QLQ-C30 is a questionnaire including 30 questions that rate the overall quality of life in cancer participants. The first 28 questions use a 4-point scale (1=not at all to 4=very much) for evaluating function (physical, role, social, cognitive, emotional), symptoms (diarrhea, fatigue, dyspnea, appetite loss, insomnia, nausea/vomiting, constipation, and pain) and financial difficulties. The last 2 questions use a 7-point scale (1=very poor to 7=excellent) to evaluate overall health and quality of life. Scores are transformed to a range of 0 to 100 using a standard EORTC algorithm. For the overall HRQoL and functioning scales, a higher score is correlated with better HRQoL, whereas a higher score represents worse HRQoL for symptom scales. Data for this outcome measure will be reported after study completion (anticipated study completion date is March 2026)
Time Frame: Up to approximately 69 months
Reporting Status: Not Posted, anticipated posting 2027-03

9. Secondary Outcome: HRQoL Assessed by European Quality of Life (EuroQol) Five-Dimensional, 3-Level (EQ-5D-3L) Score
Description: EQ-5D-3L is a health profile questionnaire consisting of the EQ-5D descriptive system and the EuroQol visual analog scale (EQ-VAS). For the EQ-5D, participants rate 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) at 1 of 3 levels (1=no problems; 2=some problems; 3=extreme problems). The EQ-5D Health Utilities Index (HUI) is derived from the five dimensions of the EQ-5D, using country-specific preference weights (tariffs) to summarize how good or bad each health state is on a scale from 1 (full health) to <0 (worse health/dead). The EQ-VAS measures self-rated global health status using a vertically oriented VAS, where 100 represents the "best imaginable health state" and 0 represents the "worst imaginable health state." Data for this outcome measure will be reported after study completion (anticipated study completion date is March 2026)
Time Frame: Up to approximately 69 months
Reporting Status: Not Posted, anticipated posting 2027-03

10. Secondary Outcome: PFS on Next-line of Therapy (PFS2)
Description: PFS2 is defined as the time from randomization to disease progression as assessed by investigator on next-line treatment or death from any cause (whichever occurred first). Data for this outcome measure will be reported after study completion (anticipated study completion date is March 2026)
Time Frame: Up to approximately 69 months
Reporting Status: Not Posted, anticipated posting 2027-03

11. Secondary Outcome: PFS by Investigator Assessment
Description: PFS by investigator assessment is defined as the time from the date of randomization to the date of first documentation of disease progression based on the investigator assessment per RECIST 1.1 or death (whichever occurred first). Data for this outcome measure will be reported after study completion (anticipated study completion date is March 2026).
Time Frame: Up to approximately 69 months
Reporting Status: Not Posted, anticipated posting 2027-03

12. Secondary Outcome: Model-predicted Clearance for Lenvatinib and Everolimus
Description: Data for this outcome measure will be reported after study completion (anticipated study completion date is March 2026)
Time Frame: Cycles 1 and 2 Day 1; 0.5-4 hours and 6-10 hours postdose; Cycle 1 Day 15: predose and 2-12 hours postdose; Cycles 3, 4, 5 and 6 Day 1: predose (Cycle length=21 days)
Reporting Status: Not Posted, anticipated posting 2027-03

13. Secondary Outcome: Area Under the Plasma Drug Concentration-time Curve (AUC) for Lenvatinib and Everolimus
Description: Data for this outcome measure will be reported after study completion (anticipated study completion date is March 2026)
Time Frame: Cycles 1 and 2 Day 1; 0.5-4 hours and 6-10 hours postdose; Cycle 1 Day 15: predose and 2-12 hours postdose; Cycles 3, 4, 5 and 6 Day 1: predose (Cycle length = 21 days
Reporting Status: Not Posted, anticipated posting 2027-03

ADVERSE EVENTS:
Time Frame: From first dose of study drug (Baseline) up to 30 days after last dose of study drug or up to data cutoff date 28 Aug 2020 (up to approximately 46 months)
Description: Safety analysis set included all participants who received at least 1 dose of any study drug.
Arm/Group | Lenvatinib 18 mg Plus Everolimus 5 mg | Lenvatinib 20 mg Plus Pembrolizumab 200 mg | Sunitinib 50 mg
All-Cause Mortality (participants affected / at risk) | 119/355 | 78/352 | 99/340
Serious Adverse Events (participants affected / at risk) | 164/355 | 178/352 | 113/340
Other Adverse Events (participants affected / at risk) | 353/355 | 351/352 | 332/340
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib 18 mg Plus Everolimus 5 mg (N=355) | Lenvatinib 20 mg Plus Pembrolizumab 200 mg (N=352) | Sunitinib 50 mg (N=340)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 4
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Eosinophilia myalgia syndrome (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 5
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 5 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 3 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 3 | 6 | 1
Myocarditis (Cardiac disorders) | 0 | 2 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Postinfarction angina (Cardiac disorders) | 1 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 7 | 0
Hypophysitis (Endocrine disorders) | 0 | 1 | 0
Hypopituitarism (Endocrine disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 3 | 0
Secondary hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Steroid withdrawal syndrome (Endocrine disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 1
Retinal vascular occlusion (Eye disorders) | 0 | 1 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0 | 0
Vogt-Koyanagi-Harada disease (Eye disorders) | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 5 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 2 | 0
Colonic fistula (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 14 | 12 | 4
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Eosinophilic gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 2 | 1
Ileus (Gastrointestinal disorders) | 2 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Immune-mediated pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 3 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 5 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 6 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 1 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Subileus (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 10 | 10 | 3
Asthenia (General disorders) | 4 | 2 | 4
Death (General disorders) | 2 | 1 | 2
Face oedema (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 2
General physical health deterioration (General disorders) | 3 | 1 | 3
Generalised oedema (General disorders) | 1 | 0 | 0
Inadequate analgesia (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 2 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 2 | 0
Oedema (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 2 | 0 | 1
Pain (General disorders) | 2 | 2 | 1
Pyrexia (General disorders) | 4 | 6 | 7
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 5 | 2 | 1
Cholecystitis acute (Hepatobiliary disorders) | 8 | 2 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 4 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1
Abdominal infection (Infections and infestations) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 1 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0
Colonic abscess (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0
Empyema (Infections and infestations) | 1 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 1 | 0
Encephalitis viral (Infections and infestations) | 0 | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 2 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1
Infectious pleural effusion (Infections and infestations) | 2 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 1 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 1
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 2 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 15 | 7 | 6
Pneumonia influenzal (Infections and infestations) | 1 | 0 | 0
Pneumonia necrotising (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Prostatic abscess (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 2 | 1
Retroperitoneal abscess (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 3 | 3
Septic arthritis staphylococcal (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Subdiaphragmatic abscess (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 4 | 4
Urosepsis (Infections and infestations) | 2 | 2 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radiation injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radiation proctitis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 2
Blood calcium increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 2
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 1
Electrocardiogram change (Investigations) | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 1
Haemoglobin increased (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 4 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 1 | 0
Transaminases increased (Investigations) | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 2 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 1 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 5 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 4
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 3 | 6 | 2
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
External ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Metastases to chest wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2 | 0
Cytotoxic oedema (Nervous system disorders) | 1 | 0 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 2 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 2
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Myasthenic syndrome (Nervous system disorders) | 0 | 1 | 0
Noninfective encephalitis (Nervous system disorders) | 0 | 1 | 0
Paralysis (Nervous system disorders) | 0 | 0 | 1
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 0 | 0 | 1
Paraparesis (Nervous system disorders) | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 2 | 1
Seizure (Nervous system disorders) | 0 | 0 | 2
Somnolence (Nervous system disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 2 | 1 | 2
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 2 | 0
Device deposit issue (Product Issues) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 2 | 0
Mania (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 5 | 0
Acute kidney injury (Renal and urinary disorders) | 10 | 8 | 5
Haematuria (Renal and urinary disorders) | 0 | 0 | 4
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 1 | 0
Nephritis (Renal and urinary disorders) | 0 | 3 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 4 | 2
Renal haemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 2 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 5
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 9 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 3
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Spinal laminectomy (Surgical and medical procedures) | 1 | 0 | 0
Aneurysm ruptured (Vascular disorders) | 0 | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 1
Embolism venous (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 8 | 2
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 2
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis migrans (Vascular disorders) | 0 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib 18 mg Plus Everolimus 5 mg (N=355) | Lenvatinib 20 mg Plus Pembrolizumab 200 mg (N=352) | Sunitinib 50 mg (N=340)
Diarrhoea (Gastrointestinal disorders) | 233 | 214 | 166
Stomatitis (Gastrointestinal disorders) | 169 | 122 | 131
Nausea (Gastrointestinal disorders) | 139 | 125 | 113
Vomiting (Gastrointestinal disorders) | 107 | 91 | 67
Constipation (Gastrointestinal disorders) | 73 | 87 | 64
Abdominal pain (Gastrointestinal disorders) | 72 | 72 | 28
Dyspepsia (Gastrointestinal disorders) | 34 | 39 | 55
Abdominal pain upper (Gastrointestinal disorders) | 45 | 34 | 26
Dry mouth (Gastrointestinal disorders) | 23 | 36 | 11
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 16 | 16 | 30
Toothache (Gastrointestinal disorders) | 24 | 19 | 9
Haemorrhoids (Gastrointestinal disorders) | 19 | 20 | 11
Abdominal discomfort (Gastrointestinal disorders) | 19 | 8 | 8
Fatigue (General disorders) | 149 | 141 | 124
Asthenia (General disorders) | 63 | 77 | 61
Oedema peripheral (General disorders) | 72 | 42 | 35
Pyrexia (General disorders) | 44 | 48 | 41
Weight decreased (Investigations) | 116 | 105 | 31
Platelet count decreased (Investigations) | 59 | 21 | 61
Lipase increased (Investigations) | 22 | 64 | 44
Aspartate aminotransferase increased (Investigations) | 52 | 39 | 37
Alanine aminotransferase increased (Investigations) | 49 | 42 | 35
Blood creatinine increased (Investigations) | 36 | 48 | 34
Amylase increased (Investigations) | 16 | 62 | 28
Blood thyroid stimulating hormone increased (Investigations) | 22 | 39 | 21
Blood cholesterol increased (Investigations) | 41 | 24 | 14
Neutrophil count decreased (Investigations) | 14 | 7 | 40
Blood triglycerides increased (Investigations) | 21 | 22 | 15
White blood cell count decreased (Investigations) | 11 | 9 | 33
Blood creatine phosphokinase increased (Investigations) | 19 | 14 | 17
Electrocardiogram QT prolonged (Investigations) | 15 | 22 | 13
Blood alkaline phosphatase increased (Investigations) | 20 | 17 | 9
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 81 | 101 | 127
Rash (Skin and subcutaneous tissue disorders) | 87 | 95 | 47
Pruritus (Skin and subcutaneous tissue disorders) | 47 | 58 | 26
Dry skin (Skin and subcutaneous tissue disorders) | 31 | 22 | 27
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 23 | 28 | 7
Yellow skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 32
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 23 | 5 | 3
Decreased appetite (Metabolism and nutrition disorders) | 143 | 142 | 105
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 80 | 42 | 41
Hypercholesterolaemia (Metabolism and nutrition disorders) | 37 | 31 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 31 | 24 | 18
Hypophosphataemia (Metabolism and nutrition disorders) | 32 | 22 | 15
Hyponatraemia (Metabolism and nutrition disorders) | 17 | 27 | 20
Hypokalaemia (Metabolism and nutrition disorders) | 30 | 22 | 11
Hyperkalaemia (Metabolism and nutrition disorders) | 14 | 27 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 75 | 99 | 52
Back pain (Musculoskeletal and connective tissue disorders) | 60 | 57 | 52
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 39 | 48 | 21
Pain in extremity (Musculoskeletal and connective tissue disorders) | 33 | 41 | 33
Myalgia (Musculoskeletal and connective tissue disorders) | 34 | 56 | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 | 24 | 12
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 20 | 16 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 84 | 70 | 53
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 84 | 105 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 50 | 51 | 32
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 70 | 25 | 37
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 33 | 23 | 12
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 19 | 12 | 0
Hypertension (Vascular disorders) | 162 | 194 | 141
Hypotension (Vascular disorders) | 17 | 24 | 6
Nasopharyngitis (Infections and infestations) | 34 | 40 | 25
Urinary tract infection (Infections and infestations) | 32 | 24 | 23
Sinusitis (Infections and infestations) | 14 | 19 | 6
Headache (Nervous system disorders) | 81 | 80 | 54
Dysgeusia (Nervous system disorders) | 59 | 42 | 95
Dizziness (Nervous system disorders) | 17 | 34 | 29
Haematuria (Renal and urinary disorders) | 15 | 17 | 19
Hypothyroidism (Endocrine disorders) | 95 | 164 | 90
Hyperthyroidism (Endocrine disorders) | 9 | 28 | 12
Anaemia (Blood and lymphatic system disorders) | 57 | 43 | 66
Thrombocytopenia (Blood and lymphatic system disorders) | 39 | 14 | 53
Neutropenia (Blood and lymphatic system disorders) | 11 | 9 | 46
Leukopenia (Blood and lymphatic system disorders) | 4 | 5 | 23
Insomnia (Psychiatric disorders) | 40 | 38 | 21
Hypomagnesaemia (Metabolism and nutrition disorders) | 17 | 27 | 13
Upper respiratory tract infection (Infections and infestations) | 24 | 31 | 21
Proteinuria (Renal and urinary disorders) | 121 | 104 | 43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT02811861/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT02811861/SAP_001.pdf